CLINICAL TRIAL: NCT05987267
Title: Nurse-led Multidisciplinary Precision Care for Patients With Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Xiuxian Zhu, Principal Investigator, Zhongshan People's Hospital, Guangdong, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K2019-017
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Nurse's Role; Multidisciplinary Communication; Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multidisciplinary precision care group (Experimental): Give the intervention of nurse-led multidisciplinary precision care
  Interventions: Other: multidisciplinary precision care
- control group (No Intervention): standard care according to guidelines

INTERVENTIONS:
Other: multidisciplinary precision care — The experimental group received precision nursing based on a multidisciplinary collaborative team in addition to standard treatment and care
  Arms: multidisciplinary precision care group

SUMMARY:
This study aimed to evaluate the feasibility and effectiveness of a nurse-led multidisciplinary precision care in early cardiac rehabilitation of patients with chronic heart failure, and further to promote the application of nurse-led multidisciplinary precision care.

DETAILED DESCRIPTION:
Enrolled patients were randomly divided as 1:1 ratio to experimental group and control group, while experimental group received nurse-led multidisciplinary precision care and the control group received standard care according to guidelines. The primary and secondary outcomes were evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years;
* Conscious, with normal cognitive function and being communicable;
* NYHA heart function class II-IV;
* Patients met the diagnostic criteria of the clinical guidelines for the diagnosis and treatment of heart failure and were diagnosed with chronic heart failure;
* Informed consent was obtained.

Exclusion Criteria:

* Patients with congenital heart disease, cardiac shock, or persistent hypotension;
* Patients with severe liver and kidney dysfunction, moderate to severe anemia or coagulation disorders, and other serious systemic complications;
* Patients with a history of mental illness, a state of severe anxiety or depression, cognitive or communication impairments, and inability to communicate and respond to investigations;
* Patients have been involved in other research that would interfere with this study;
* Patients who declined cardiac rehabilitation and signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction | baseline, pre-intervention, 1 month after intervention, 3 months after intervention
6-minute walking distance | baseline, pre-intervention, 1 month after intervention, 3 months after intervention

SECONDARY OUTCOMES:
the European Organization for Research and Treatment of Cancer (EORTC) quality-of-life (QoL) questionnaires (QLQ) QLQ-C30 (version 3.0) score Quality of Life | baseline, pre-intervention, 1 month after intervention, 3 months after intervention
Symptom Check List-90 | baseline, pre-intervention, 1 month after intervention, 3 months after intervention
Performance Status Score | baseline, pre-intervention, 1 month after intervention, 3 months after intervention
Numbers of patients with cardiovascular complications | baseline, pre-intervention, 1 month after intervention, 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Xiuxian Zhu, Study Chair — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No